CLINICAL TRIAL: NCT06316752
Title: The Natural History of Sialidosis Type I
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Professor, National Taiwan University Hospital
Other Study IDs: 202107158RINB
Record Dates: First submitted 2024-02-26; First posted 2024-03-18 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Observational Study
Keywords: sialidosis; NEU1 gene; Natural history
MeSH Terms: conditions — Mucolipidoses | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A maximum of 10ml of blood will be drawn from recruited patient. DNA will be extracted and the plasma will be retained for possible use in the future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with sialidosis type 1: Patients with a definite diagnosis of this disease are candidates for this study.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — It is an observational study involving non-invasive routine examinations without treatment, thus posing no additional risk to patients. This project does not involve the use of medications, medical techniques, or the market status of medical equipment.

SUMMARY:
Sialidosis type 1 is an autosomal recessive disorder caused by bialleic NEU1 gene mutations. Patients with sialidosis type I present variable neurological and eye dysfunction and the progression rate is variable. The goal of this protocol is to assess the neurological and ophthalmological status of these patients and characterize the clinical and laboratory abnormalities in order to determine the natural history of the disease. Patients will be followed every 6 month with comprehensive clinical, neurological and ophthalmological examinations combined with neuropsychological, blood, radiological and electrophysiological tests.

DETAILED DESCRIPTION:
Sialidosis is a rare autosomal recessive genetic disorder caused by a deficiency of sialidase with an estimated prevalence rate of one patient per 250,000 people. Sialidase, also known as neuraminidase I or NEU1, is an enzyme found inside lysosomes. Patients with sialidosis lack NEU1 due to genetic mutations, leading to low levels or impaired function of sialidase in cells. As a result, sialic acid cannot be effectively removed from glycoproteins or glycolipids, causing abnormal accumulation of these substances in cells, which can lead to cellular dysfunction or even death. Sialidosis is divided into two types: Type II patients show severe symptoms in infancy, while Type I patients develop symptoms from childhood to adolescence, followed by a slow, progressive deterioration. Typical symptoms of Type I sialidosis begin with unsteady gait and may include progressive visual impairment, muscle twitches (myoclonus), muscle weakness and atrophy, coordination difficulties, seizures, and mild intellectual disability. As muscle tremors worsen, activities like sitting, standing, and walking become challenging. Progressive vision loss can cause color blindness or night blindness, and cherry-red spot abnormalities may appear on eye exams.

The progressive nature of the Sialidosis type is variable. Some patients have clear deterioration, while others seem to stay at the same level of the disease for a long time. This study aims to track the natural history of patients with sialidosis type I to identify suitable clinical markers for measuring disease progression speed. It is an observational study involving non-invasive routine examinations without treatment, thus posing no additional risk to patients.

Patients with a definite diagnosis of this disease are candidates for this study. Patients will receive physical and neurological examination every 6 month with a total duration of 24 months. A history will be taken and a physical exam done. Blood and urine tests will be done along with brain wave recording, complete eye examination, cognitive test, gait analysis, and myoclonus evaluation. A maximum of 10ml of blood will be drawn from recruited patient. Various eye tests will also be done. DNA will be extracted and the plasma will be retained for possible use in the future studies. Brain MRI without contrast, evoked potentials of visual and somatosensory systems, nerve conduction study and nerve excitability test will be done annually. Medication record and the response to treatment will be recorded as well. There is a possibility of improved medical management and rehabilitative treatment as a result of participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must:

  * Genetic diagnosis of sialidosis type I
  * Able to tolerate a general exam and neurological exam
  * Able to tolerate a modest amount of blood drawing
  * Able to tolerate the complete electrophysiological studies
  * Able to tolerate the performance of electroencephalogram and brain MRI
  * Able to tolerate a neuropsychological testing and opathalmology evaluation

Exclusion Criteria:

* Patients who cannot tolerate the scheduled examinations and blood drawing

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patieints who have a definitive diagnosis of sialidosis type I based on genetic test
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | every 6 months up to 1 year
  SARA is a clinical scale that is based on a semi-quantitative assessment of cerebellar ataxia on an impairment level. It can also be used as a rehabilitation index of gait status and ADL independence in ataxic patients. The range of SARA scre is 0-40. The higer score means the worse status.
Unified Myoclonus Rating Scale (UMRS) | every 6 months up to 1 year
  The UMRS score for each task is a multiplied measure of the myoclonus amplitude and frequency of the participant. The range of UMRS is 0-128. The higer score means the worse status.

SECONDARY OUTCOMES:
MRI of the brain | every 1 year
  brain structure evaluation using T2 weighted images on 3T scanner
Blood test for alpha-N -acetyl neuraminidase activity and neruofilamment light chain | every year
  Blood biomarkers to reflect the disease severity of the disease progression
Electrophysyiology test on peripheral nerves | every year
  Evaluate the peripheral nerve conduction velocity.
Opathalmology examinations for cherry-red spots | every year
  Evaluate the existence of cherry red spot
Montreal cognitive assessment score | every year
  Evaluate the cognitive function (the higher score means the better cognitive function)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan